CLINICAL TRIAL: NCT01182740
Title: Comparison of Endotracheal Intubation Success Rates Using Video Laryngoscopes in Entrapped Patients - a Manikin Study
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Responsible Party: Wolfgang A. Wetsch, M.D., Department of Anaesthesiology, University Hospital of Cologne, Germany
Other Study IDs: 10-183
Record Dates: First submitted 2010-08-13; First posted 2010-08-17 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2010-08

CONDITIONS: Endotracheal Intubation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- glidescope
- storz c-mac
- mcgrath vl
- ambu pentax aws
- macintosh laryngoscope
- others

SUMMARY:
The investigators will compare the success rates of endotracheal intubation in a simulated entrapped car accident victim (manikin) using different video laryngoscopes by experienced emergency physicians.

The investigators hypothesized that video laryngoscopes may improve success rates.

ELIGIBILITY:
Inclusion Criteria:

* experienced emergency physicians

Exclusion Criteria:

* no experience in out-of-hospital emergency medicine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: experienced emergency physicians
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-08; Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
successful endotracheal intubation | 2 months
  We compare the success rates of endotracheal intubation with the different devices

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Cologne, Cologne, Germany

REFERENCES:
- [Derived] Wetsch WA, Carlitscheck M, Spelten O, Teschendorf P, Hellmich M, Genzwurker HV, Hinkelbein J. Success rates and endotracheal tube insertion times of experienced emergency physicians using five video laryngoscopes: a randomised trial in a simulated trapped car accident victim. Eur J Anaesthesiol. 2011 Dec;28(12):849-58. doi: 10.1097/EJA.0b013e32834c7c7f. PMID 21986981